CLINICAL TRIAL: NCT01718262
Title: Study Measuring Total Plasma Ropivacaine Levels During Continuous Peripheral Nerve Catheter Infusion
Status: Completed | Type: Observational
Sponsor: Defense and Veterans Center for Integrative Pain Management (Other)
Responsible Party: Sponsor
Other Study IDs: 353368-19
Record Dates: First submitted 2012-10-17; First posted 2012-10-31 (Estimated); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Anesthesia
Keywords: Ropivacaine Level; continuous peripheral nerve blocks.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The plasma ropivacaine samples will be assayed at the Department of Research Programs Laboratory (DRP) at WRNMMC. Once the whole blood sample has been centrifuged, the plasma will be removed with a glass pipette, placed in a storage container. The blood samples will be labeled with a non sequential serial number and will not include the time of the blood draw. This will blind the DRP laboratory to the patient's identity and timing of the blood draw.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to measure the blood levels of the medicine called ropivacaine (local anesthetic) used to manage pain. Ropivacaine is a widely used medication and is not the subject of this study, but the investigators are studying how much of the drug can be found in the patient's blood, known as the blood level, of this medicine. Too much ropivacaine in a patient's blood can lead to local anesthetic toxicity. Once the nerve catheter is removed, local anesthetic toxicity is no longer a potential problem. However, there is little data on what ropivacaine blood levels are after having the catheter in for a long period of time(up to one month).

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years and older, capable of providing informed consent indicating awareness of the investigational nature of the study, in keeping with institutional policy
* Written informed consent must be obtained from each patient prior to entering the study
* Patients must be scheduled to receive a continuous peripheral nerve catheter

Exclusion Criteria:

* Refusal to have serial blood drawn
* Contraindication for a continuous peripheral nerve catheter (allergy to local anesthetic, infection at site of injection, elevated coagulation times (international normalized ratio (INR)>1.5, partial thromboplastin time (PTT)>38; these values are drawn as part of routine standard of care and those values will be checked prior to initial catheter insertion), therapeutic dosing of anticoagulation medication, moderate to severe head injury and moderate to severe traumatic brain injury
* Patients with a hematocrit < 20. Complete Blood Counts (CBCs) are drawn as part of routine standard of care and will be followed by the Acute Pain Service. Although the CBCs and ropivacaine blood draws will not always coincide, we will always check the last hematocrit obtained prior to our blood draw
* Severe liver or renal disease (values greater than two times normal range)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Military health care beneficiaries age 18 years and older presenting for upper or lower extremity surgery requiring continuous infusions of local anesthetic either at WRNMMC will be asked to participate in the study. We will recruit up to fifty patients for the study at WRNMMC.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2010-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Plasma Ropivicaine Levels | up to 10 days
  Blood will be drawn every 0, 3, 5, 7, and 10 days. Blood is drawn every 3 days thereafter.

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States